CLINICAL TRIAL: NCT01907854
Title: Efficacy and Safety of Switching From Sitagliptin to Liraglutide in Subjects With Type 2 Diabetes Not Achieving Adequate Glycaemic Control on Sitagliptin and Metformin
Acronym: LIRA-SWITCH™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-4059; 2012-004931-22 (EudraCT Number); U1111-1136-2073 (Other: WHO); CTRI/2014/05/004623 (Registry Identifier: Clinical Trial Registry India (CTRI))
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Results first posted 2016-07-01 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide + metformin + sitagliptin placebo (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo
- Sitagliptin + metformin + liraglutide placebo (Experimental)
  Interventions: Drug: sitagliptin; Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Starting dose of 0.6 mg/day, with weekly dose escalations of 0.6 mg/day until the maintenance dose of 1.8 mg/day is reached. Administered subcutaneously (s.c., under the skin) once daily + metformin tablets (at least 1000 mg/day)
  Arms: Liraglutide + metformin + sitagliptin placebo
Drug: sitagliptin — 100 mg/day sitagliptin tablets once-daily + metformin (at least 1000 mg/day)
  Arms: Sitagliptin + metformin + liraglutide placebo
Drug: placebo — Sitagliptin placebo tablets once-daily
  Arms: Liraglutide + metformin + sitagliptin placebo
Drug: placebo — Sitagliptin placebo tablets once-daily
  Arms: Sitagliptin + metformin + liraglutide placebo

SUMMARY:
This trial is conducted in Asia, Europe and North America. The aim of the trial is to investigate the efficacy and safety of switching from sitagliptin to liraglutide in subjects with type 2 diabetes not achieving adequate glycaemic control on sitagliptin and metformin.

ELIGIBILITY:
Inclusion Criteria:

* - Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* - Subjects diagnosed with type 2 diabetes and treated with metformin equal to or above 1500 mg/day (or maximum tolerated dose equal to or above 1000 mg/day) and sitagliptin 100 mg/day, both at a stable dose for at least 90 days prior to screening. Stable is defined as unchanged medication and dose
* - HbA1c 7.5% - 9.5% (58 mmol/mol - 80 mmol/mol) (both inclusive)
* - Body mass index equal to or above 20 kg/m^2

Exclusion Criteria:

* - Any chronic disorder or severe disease which at the discretion of the investigator might jeopardise subject's safety or compliance with the protocol
* - Treatment with glucose lowering agent(s) other than stated in the inclusion criteria in a period of 90 days prior to screening. An exception is short-term treatment (equal to or less than 7 days in total) with insulin in connection with intercurrent illness
* - Female who is pregnant, breast-feeding, intends to become pregnant or of child-bearing potential not using adequate contraceptive methods (adequate contraceptive measures as required by local regulations or practice)
* - History of chronic pancreatitis or idiopathic acute pancreatitis
* - Screening calcitonin value equal to or above 50 ng/L
* - Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
* - Diagnosis of malignant neoplasm in the previous 5 years (except basal cell skin cancer or squamous cell skin cancer)
* - Impaired liver function, defined as alanine aminotransferase equal to or above 2.5 times upper normal limit
* - Impaired renal function defined as estimated glomerular filtration rate 60 mL/min/1.73 m^2 per modification of diet in renal disease formula
* - Any episode of unstable angina, acute coronary event, cerebral stroke/transient ischemic attack or other significant cardiovascular event as judged by the investigator within 90 days prior to screening
* - Heart failure, New York Heart Association class IV
* - Uncontrolled treated or untreated hypertension (systolic blood pressure equal to or above 180 mmHg and/or diastolic blood pressure equal to or above 100 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2013-12-02 (Actual); Primary Completion 2015-06-15 (Actual); Study Completion 2015-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (93):
- United States (49):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Mission Viejo, California
  - Novo Nordisk Investigational Site, Roseville, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Chiefland, Florida
  - Novo Nordisk Investigational Site, Fort Lauderdale, Florida
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, North Miami, Florida
  - Novo Nordisk Investigational Site, Port Charlotte, Florida
  - Novo Nordisk Investigational Site, Johns Creek, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Blackfoot, Idaho
  - Novo Nordisk Investigational Site, Arlington Heights, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Skokie, Illinois
  - Novo Nordisk Investigational Site, Avon, Indiana
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Council Bluffs, Iowa
  - Novo Nordisk Investigational Site, Bangor, Maine
  - Novo Nordisk Investigational Site, Fall River, Massachusetts
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, City of Saint Peters, Missouri
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Elizabeth, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Salisbury, North Carolina
  - Novo Nordisk Investigational Site, Akron, Ohio
  - Novo Nordisk Investigational Site, Reading, Pennsylvania
  - Novo Nordisk Investigational Site, Moncks Corner, South Carolina
  - Novo Nordisk Investigational Site, Orangeburg, South Carolina
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Edinburg, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, New Braunfels, Texas
  - Novo Nordisk Investigational Site, North Richland Hills, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Virginia Beach, Virginia
  - Novo Nordisk Investigational Site, Spokane, Washington
- Canada (15):
  - Novo Nordisk Investigational Site, Surrey, British Columbia
  - Novo Nordisk Investigational Site, Brampton, Ontario
  - Novo Nordisk Investigational Site, Burlington, Ontario
  - Novo Nordisk Investigational Site, Concord, Ontario
  - Novo Nordisk Investigational Site, Etobicoke, Ontario
  - Novo Nordisk Investigational Site, Grimsby, Ontario
  - Novo Nordisk Investigational Site, Ottawa, Ontario
  - Novo Nordisk Investigational Site, Sarnia, Ontario
  - Novo Nordisk Investigational Site, Strathroy, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Drummondville, Quebec
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Saint Romuald, Quebec
  - Novo Nordisk Investigational Site, Trois-Rivières, Quebec
  - Novo Nordisk Investigational Site, Québec
- Hungary (8):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Eger
  - Novo Nordisk Investigational Site, Gyula
  - Novo Nordisk Investigational Site, Salgótarján
  - Novo Nordisk Investigational Site, Sopron
  - Novo Nordisk Investigational Site, Szeged
  - Novo Nordisk Investigational Site, Tatabánya
- India (8):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Visakhapatnam, Andhra Pradesh
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Gandhinagar, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, New Delhi
- Israel (6):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Herzliya
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Nahariya
  - Novo Nordisk Investigational Site, Ofakim
  - Novo Nordisk Investigational Site, Tel Aviv
- Novo Nordisk Investigational Site, San Juan, Puerto Rico
- Spain (6):
  - Novo Nordisk Investigational Site, Badalona
  - Novo Nordisk Investigational Site, Ferrol
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Sanlúcar de Barrameda
  - Novo Nordisk Investigational Site, Seville

REFERENCES:
- [Result] Bailey TS, Takacs R, Tinahones FJ, Rao PV, Tsoukas GM, Thomsen AB, Kaltoft MS, Maislos M. Efficacy and safety of switching from sitagliptin to liraglutide in subjects with type 2 diabetes (LIRA-SWITCH): a randomized, double-blind, double-dummy, active-controlled 26-week trial. Diabetes Obes Metab. 2016 Dec;18(12):1191-1198. doi: 10.1111/dom.12736. Epub 2016 Sep 14. PMID 27381275
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 86 sites in 6 countries: Canada (14); Hungary (8); India (7); Israel (8); Spain (6); and United States (43).
Pre-assignment Details: Screening details: Subjects were adult males or females with type 2 diabetes mellitus (T2DM) who had inadequate glycaemic control with stable doses of sitagliptin and metformin for 90 days prior to screening.
Groups:
- Liraglutide: Subjects in this arm received treatments for a duration of 26 weeks; once-daily (OD) liraglutide (s.c., [under the skin] injection 0.6 mg/day, with weekly dose escalations of 0.6 mg/day up to a maintenance dose of 1.8 mg/day) + metformin tablets (≥1500 mg/day [or documented maximum tolerated dose
  ≥1000 mg/day]) + OD sitagliptin placebo tablets.
- Sitagliptin: Subjects in this arm received treatments for a duration of 26 weeks; OD sitagliptin tablets (100 mg) + metformin tablets (≥1500 mg/day [or documented maximum tolerated dose ≥1000 mg/day]) + OD s.c., injection of liraglutide placebo.
Period: Overall Study
Arm/Group | Liraglutide | Sitagliptin
Started | 203 | 204
Exposed | 202 (One subject in lira arm was not exposed (Reason: withdrawal by subject)) | 204
Completed | 187 | 191
Not Completed | 16 | 13
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Lost to Follow-up | 2 | 2
Not completed — Unclassified | 4 | 3

BASELINE CHARACTERISTICS:
Population: Demographics and baseline characteristics of all exposed subjects are summarised in continuous variables. There were missing baseline values for fasting plasma glucose in 2 subjects in the liraglutide arm and 1 subject in the sitagliptin arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Sitagliptin | Total
Number analyzed (Participants) | 202 | 204 | 406
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.6) | 56.5 (9.7) | 56.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 79 | 164
  Male | 117 | 125 | 242
HbA1c [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.3 (0.6) | 8.2 (0.6) | 8.3 (0.6)
Body Weight [Mean (Standard Deviation); unit: kg] | 88.9 (19.8) | 91.2 (19.6) | 90.1 (19.7)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mmol/L] | 10.0 (2.7) | 9.7 (2.5) | 9.9 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin)
Description: Change from baseline in HbA1c was analysed after 26 weeks of treatment. Analysis population set: full analysis set (FAS); all randomised subjects receiving at least one dose of any of the trial products. Missing values were imputed using mixed model for repeated measurements (MMRM).
Time Frame: From baseline to week 26
Population: Full analysis set (FAS) -All randomised subjects receiving at least one dose of any of the trial product.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | Liraglutide | Sitagliptin
Number analyzed (Participants) | 176 | 182
percentage of glycosylated haemoglobin | -1.146 (0.9748) | -0.529 (1.0148)
Statistical Analysis 1: Comparison: Liraglutide vs Sitagliptin; Changes in HbA1c from baseline to the 26 weeks measurements were analysed using MMRM, with treatment, baseline HbA1c level (≤8.5% and >8.5%), metformin dose (<1500 mg/day and ≥1500 mg/day), the interaction between baseline HbA1c level and metformin dose, and country as factors and the HbA1c value at baseline as a covariate, all variables nested within week as a factor; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Superiority of liraglutide over sitagliptin was concluded if the 95% Confidence Interval for the treatment difference was entirely below 0%; Treatment difference = -0.61, 95% CI 2-sided [-0.82 to -0.40]

2. Secondary Outcome: Change in Body Weight
Description: Change from baseline in body weight was analysed after 26 weeks of treatment. Analysis population set: FAS: all randomised subjects receiving at least one dose of any of the trial products. Missing values were imputed using MMRM.
Time Frame: From baseline to week 26
Population: FAS - All randomised subjects receiving at least one dose of any of the trial product.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide | Sitagliptin
Number analyzed (Participants) | 192 | 200
kg | -3.32 (3.135) | -1.80 (2.974)
Statistical Analysis 1: Comparison: Liraglutide vs Sitagliptin; Change in body weight from baseline to the 26 weeks measurements was analysed using MMRM, with treatment, baseline HbA1c level (≤8.5% and >8.5%), metformin dose (<1500 mg/day and ≥1500 mg/day), the interaction between baseline HbA1c level and metformin dose, and country as factors and the body weight at baseline as a covariate and all variables nested within week as a factor; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Treatment difference = -1.67, 95% CI 2-sided [-2.34 to -0.99]

3. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change from baseline in fasting plasma glucose was analysed after 26 weeks of treatment. Missing values were imputed using MMRM.
Time Frame: From baseline to week 26
Population: FAS - All randomised subjects receiving at least one dose of any of the trial product.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Liraglutide | Sitagliptin
Number analyzed (Participants) | 190 | 199
nmol/L | -1.967 (2.3585) | -0.588 (2.1363)

4. Secondary Outcome: Change in Fasting Blood Lipids
Description: Ratio to baseline in fasting blood lipids (total cholesterol, low density lipoprotein [LDL], very low density lipoprotein [VLDL], high density lipoprotein [HDL], triglycerides, and free fatty acids) were analysed after 26 weeks treatment. Missing values were imputed using MMRM. Here we are presenting ratio to baseline data.
Time Frame: From baseline to week 26
Population: FAS-All randomised subjects receiving at least one dose of any of the trial product. There were missing baseline values for free fatty acids in 1 subject in the liraglutide arm and 6 subjects in the sitagliptin arm.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Liraglutide | Sitagliptin
Number analyzed (Participants) | 155 | 156
ratio
  Total cholesterol | 1.011 (0.1906) | 1.045 (0.2323)
  LDL cholesterol | 1.049 (0.3899) | 1.121 (0.4661)
  VLDL cholesterol | 1.062 (0.4236) | 1.075 (0.4625)
  HDL cholesterol | 1.004 (0.1528) | 0.997 (0.1548)
  Triglycerides | 1.089 (0.4975) | 1.099 (0.4889)
  Free Fatty acids | 1.086 (0.774) | 1.104 (0.5839)

5. Secondary Outcome: Change in Systolic Blood Pressure and Diastolic Blood Pressure
Description: Change from baseline in systolic and diastolic blood pressure were analysed after 26 weeks of treatment. Missing values were imputed using MMRM.
Time Frame: From baseline to week 26
Population: FAS - All randomised subjects receiving at least one dose of any of the trial product
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liraglutide | Sitagliptin
Number analyzed (Participants) | 192 | 200
mmHg
  Systolic Blood Pressure | -3.6 (11.596) | -2.57 (11.593)
  Diastolic Blood Pressure | -0.23 (7.085) | -0.81 (7.193)

6. Secondary Outcome: Subjects Who Achieve HbA1c Below 7.0% (53 mmol/Mol) (American Diabetes Association Target) (y/n)
Description: Number of subjects who achieve HbA1c <7.0% were analysed after 26 weeks of treatment. Missing values were imputed using MMRM.
Time Frame: After 26 weeks of treatment
Population: FAS-All randomised subjects receiving at least one dose of any of the trial product.
Measure: Number; unit: percentage (%)
Arm/Group | Liraglutide | Sitagliptin
Number analyzed (Participants) | 176 | 182
percentage (%)
  Yes | 50.6 | 26.9
  No | 49.4 | 73.1

7. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: A treatment emergent adverse event (TEAE) was defined as an event that had an onset date (or increase in severity) on or after the first day of exposure to randomised treatment and no later than seven days after the last day of randomised treatment. The number of TEAEs was recorded during 26 weeks of treatment plus one week follow-up period.
Time Frame: During 26 weeks of treatment plus one week follow-up period.
Population: Safety analysis set-All randomised subjects receiving at least one dose of any of the trial product.
Measure: Number; unit: number of events
Arm/Group | Liraglutide | Sitagliptin
Number analyzed (Participants) | 202 | 204
number of events | 455 | 318

ADVERSE EVENTS:
Time Frame: 27 weeks (26 weeks of treatment period + 1 week of follow-up)
Description: Adverse events were collected for safety analysis set that included all subjects who received at least one dose of any of the trial products.
Arm/Group | Liraglutide | Sitagliptin
Serious Adverse Events (participants affected / at risk) | 6/202 | 7/204
Other Adverse Events (participants affected / at risk) | 96/202 | 61/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=202) | Sitagliptin (N=204)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=202) | Sitagliptin (N=204)
Diarrhoea (Gastrointestinal disorders) | 33 (45) | 19 (21)
Nausea (Gastrointestinal disorders) | 44 (59) | 16 (21)
Vomiting (Gastrointestinal disorders) | 15 (18) | 10 (15)
Nasopharyngitis (Infections and infestations) | 12 (14) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 12 (12) | 13 (15)
Lipase increased (Investigations) | 11 (12) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 18 (18) | 7 (7)
Headache (Nervous system disorders) | 13 (16) | 12 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more public disclosures may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property. The results of this trial will be subject to public disclosure on external web sites according to international regulations, as reflected in the Novo Nordisk Code of Conduct for Clinical Trial Disclosure.